CLINICAL TRIAL: NCT03888898
Title: Just-in-time Elastomeric Training and Fit Testing (JET FIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Emory University (Other); The University of Texas Health Science Center, Houston (Other); Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Elastomeric Base Protocol
Record Dates: First submitted 2019-03-11; First posted 2019-03-25 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Infection
Keywords: N95 filtering facepiece respirators; elastomeric respirators; public health emergency; healthcare workers; occupational health; respiratory protection program; personal protective equipment; airborne transmissible pathogens; reusable respirator
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N95 Filtering Facepiece Respirator (Active Comparator): control fit testing
  Interventions: Other: Control fit test evaluation
- Elastomeric Respirator (Experimental): experimental rapid conversion fit testing and competency evaluations
  Interventions: Other: Reusable respirator fit test and competency evaluation

INTERVENTIONS:
Other: Reusable respirator fit test and competency evaluation — Feasibility of rapid conversion to reusable elastomeric respirator use during public health emergency
  Arms: Elastomeric Respirator
Other: Control fit test evaluation — control comparator for fit testing time threshold
  Arms: N95 Filtering Facepiece Respirator

SUMMARY:
This is a clinical trial to evaluate feasibility of a just in time elastomeric half mask respirator (EHMR) fit test and competency training for healthcare personnel (HCP) during a simulated public health emergency.

DETAILED DESCRIPTION:
This is a national multicenter pragmatic demonstrative clinical trial to evaluate feasibility of a just in time elastomeric half mask respirator (EHMR) fit test and competency training for healthcare personnel (HCP) during a simulated public health emergency. This study will assess participant and institution ability to rapidly convert and demonstrate proficiency using reusable respirators in the healthcare field to provide a stopgap for respiratory protection program guidelines in times of disposable respirator supply shortages. This protocol is the first in a series of three studies included in the Assessment of Elastomeric Respirators in Healthcare Delivery Settings project sponsored by the National Institute for Occupational Safety and Health (NIOSH) at the Centers for Disease Control and Prevention (CDC). This project is funded in kind by the National Personal Protective Technology Laboratory (NPPTL), the Office of Public Health Preparedness and Response (OPHPR), and the National Center for Immunization and Respiratory Diseases (NCIRD). The first of three protocols, this will be followed by laboratory and field studies assessing disinfection methods and routine use EHMR. Three (3) United States (US) healthcare delivery organizations (University of Texas Houston, Wayne State University, and Emory University) will be included as study sites in this base protocol, individually accruing a participant sample size up to 100 HCP, with a minimum of 50 evaluable participants per site. A total sample size of 150 to 300 evaluable participants are expected to be accrued nationally. The purpose of this Base protocol is to assess feasibility of reusable EHMRs in healthcare for a just in time adaptation during respiratory infectious disease outbreaks, epidemics, pandemics, and/or disposable respirator supply shortages.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand, the willingness to participate, and the completion of a written informed consent document
* Understands spoken and written English language as required for consent, demonstration videos, demonstration checklist, and evaluation measures
* Age > 18 years old
* Medical Evaluation Form completed by the participant and reviewed/signed by a licensed medical professional such as a registered nurse, nurse practitioner, physician assistant, or physician
* If a subject reports "yes" to any medical condition listed on the Medical Evaluation Form in Part B Questions 2, 5, 6, and/or 7, a Physician must review the subject's current and past medical history and provide documented clearance for them to participate.
* Healthcare personnel requiring respiratory protection, included in the hospital's Respiratory Protection Program and able to provide estimated number of years using respirators
* Bivariate Panel facial measurements and completed data capture form
* Review of the General Photo Release Form. This allows photos and/or videos taken during study participation to be utilized in presentations and publications or the post study webinars contracted (photos/videos will not contain participant personal identifiers). Participants may decline completing this form (and if they decline, they may not be included in any photos or videos). Documented verification of agreement or decline must be addressed before registration to study
* Passed the Taste Threshold test with a score recorded of 10, 20, or 30, indicating participant can taste the sodium saccharin challenge agent for the qualitative fit test
* Eligibility Checklist

Exclusion Criteria:

* Inability to adhere to study and/or follow up procedures
* Facial hair or piercings, which may interfere with the facial seal region of the elastomeric respirator
* Individuals with facial deformities/injuries that may prevent seal and/or passing a fit test
* Known hypogeusia or ageusia (decreased ability to taste certain types of foods or the absence of taste entirely which precludes qualitative fit test)
* Inability to ensure availability for the study intervention date(s) selected by site personnel
* Chronic or current pulmonary or lung problems reported by subject (reports "yes" to any item in Part B. questions 3 or 4) on Medical Evaluation Form
* Prior problems using a respirator as reported in Part B. question 8 of the Medical Evaluation Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Fit test pass and fail rates in healthcare | within 2 hours
  Participant subjective pass or fail result for sodium saccharin aerosol qualitative fit test
Competency Evaluation | within 2 hours
  elastomeric half mask respirator participant "Competency Evaluation" determined by measuring competence based on tasks completed by participants using a numeric scale of 26-78 points possible. 6 competencies will be tested with subparts defined as tasks (5 competencies include 4 tasks and 1 competency includes 6 tasks). Each task is 1-3 points, with 3 points being the highest score and 1 point being the lowest possible score.

SECONDARY OUTCOMES:
User seal check predictive value | within 2 hours
  subjective pass or fail reported scores by subjects during user seal checks
Bivariate Panel facial measurement accuracy for respirator size allocations | within 60 days
  Bivariate Panel cell category allocation accuracy measured by pass or fail of fit test
Respirator fit test time threshold | within 2 hours
  Measurement of maximum time threshold for training required to convert subjects to disposable and reusable respirators

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Radonovich, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Wayne State University, Detroit, Michigan
  - University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No